CLINICAL TRIAL: NCT06343805
Title: A Multicenter, Open-Label, Phase 1 Study of AJ1-11095 Administered as Oral Monotherapy in Patients With Primary Myelofibrosis (PMF), Post-Polycythemia Vera Myelofibrosis (PPV-MF), or Post-Essential Thrombocythemia Myelofibrosis (PET-MF) Who Have Been Failed by a Type I JAK2 Inhibitor (JAK2i)
Brief Title: A Phase 1 Study of AJ1-11095 in Patients With Primary Myelofibrosis (PMF), Post-Polycythemia Vera Myelofibrosis (PPV-MF), or Post-Essential Thrombocythemia Myelofibrosis (PET-MF) Who Have Been Failed by a Type I JAK2 Inhibitor (JAK2i)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ajax Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AJX-101
Record Dates: First submitted 2024-03-13; First posted 2024-04-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Primary Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; PMF; PPV-MF; PET-MF
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Intervention Model Description: This dose escalation study will follow a 3+3 cohort design until the RP2D and/or MTD is determined.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): Dose A of AJ1-11095 taken orally by patients.
  Interventions: Drug: AJ1-11095
- Cohort 2 (Experimental): Dose B of AJ1-11095 taken orally by patients.
  Interventions: Drug: AJ1-11095
- Cohort 3 (Experimental): Dose C of AJ1-11095 taken orally by patients.
  Interventions: Drug: AJ1-11095
- Cohort 4 (Experimental): Dose D of AJ1-11095 taken orally by patients.
  Interventions: Drug: AJ1-11095
- Cohort 5 (Experimental): Dose E of AJ1-11095 taken orally by patients.
  Interventions: Drug: AJ1-11095
- Dose Expansion Cohort 1 (Experimental): Candidate RP2D of AJ1-11095 taken orally by patients.
  Interventions: Drug: AJ1-11095
- Dose Expansion Cohort 2 (Experimental): Alternative candidate RP2D of AJ1-11095 taken orally by patients.
  Interventions: Drug: AJ1-11095

INTERVENTIONS:
Drug: AJ1-11095 — Type II JAK2 Inhibitor

SUMMARY:
AJX-101 is a first-in-human (FIH), phase 1, non-randomized, multi-center, open-label clinical trial designed to investigate the safety, tolerability, pharmacokinetics (PK), clinical activity and changes in biomarkers of an orally administered type II JAK2 inhibitor, AJ1-11095, in subjects with primary or secondary myelofibrosis previously treated with at least one type I JAK2 inhibitor.

DETAILED DESCRIPTION:
This is a phase 1, non-randomized, open-label study utilizing a 3+3 sequential dose escalation design followed by an expansion phase. The primary objective will be to evaluate the safety and tolerability of AJ1-11095, and establish a Maximally Tolerated Dose (MTD) and/or inform the establishment of a candidate Recommended Phase 2 dose (RP2D). The RP2D may be the maximally tolerated dose (MTD) or may be a dose below the MTD. The candidate RP2D will be based on AE pattern, PK and biomarker information, in addition to all available safety and efficacy data. Expansion cohorts will be enrolled to gather additional safety and efficacy information and to further refine input for future RP2D discussions. Eligible participants will have PMF, PPV-MF or PET-MF and will have either have relapsed after a response, or be refractory to, at least one prior type I JAK2 inhibitor therapy, either administered as monotherapy or in combination with another drug.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Diagnosis of PMF, post-PV MF, or post-ET MF.
3. DIPSS Intermediate-2 or High-risk MF with ≤10% blasts, regardless of JAK2 mutation status.
4. Estimated spleen volume ≥450cm3.
5. MFSAF v.4.0 TSS ≥10, or at least 2 of 7 MFSAF-assessed symptoms with scores ≥3.
6. ECOG PS of 0, 1, 2, or 3.
7. Prior therapy with at least 1 type I JAK2 inhibitor, and either failed to achieve a response or relapsed after achieving a response.
8. ANC ≥1.0×10^9/L.
9. Platelet count ≥75×10^9/L.
10. eGFR ≥45 mL/min/1.73m2.
11. Serum total bilirubin ≤2.0 × upper limit of normal (ULN).
12. AST and ALT ≤3.0 × ULN.
13. QTcF ≤480 msec.

Exclusion Criteria:

1. Prior splenectomy.
2. Splenic irradiation within 3 months prior to first dose of study drug.
3. Ongoing use of systemic corticosteroids at dose equivalent to >10mg/day of prednisone.
4. Uncontrolled intercurrent illness such as an acute infection.
5. Chronic active or acute hepatitis B or C infection.
6. Chemotherapy in the previous 4 weeks prior to first dose of study drug (Hydrea is permitted until 5 days before starting protocol therapy).
7. Use of a Type I JAK2 inhibitor must have been discontinued for at least 5 days or 5 half-lives prior to dosing (whichever is longer).
8. Use of erythropoiesis stimulating agents (unless stable for >8 weeks).
9. Peripheral neuropathy ≥ Grade 2 (NCI CTCAE v 5.0).
10. Unable or unwilling to undergo CT or MRI for spleen size imaging.
11. Pregnant or breastfeeding.
12. Requirement for therapy with a medication that is a strong CYP3A4 inhibitor as a concomitant medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment-emergent adverse events as assessed by CTCAE v 5.0. | Baseline through study completion, an average of 1 year
  Treatment Emergent AEs will be assessed during routine study visits and compared to Baseline to continuously evaluate safety and tolerability of AJ1-11095.
Number of patients with Dose Limiting Toxicities (DLTs) | Baseline through study completion, an average of 1 year
  Protocol-defined potential DLTs will be assessed by the Safety Review Committee at routine intervals.
To establish the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of AJ1-11095 | Baseline through study completion, an average of 1 year
  Safety evaluations will occur consistently for each patient and across patients to assess MTD or RP2D. See description of safety evaluations described in outcomes 1 and 2 mentioned above.

SECONDARY OUTCOMES:
To assess clinical response to AJ1-11095 evaluated by the Total Symptom Score (TSS). | Baseline through Week 24
  Number and proportion of patients with an improvement of ≥50% from Baseline in Total TSS as well as time to TSS response and duration of TSS response using the Myelofibrosis Symptom Assessment Form (MFSAF) v4.0. The TSS is a 7 question assessment form with lower scores indicating better outcomes.
To assess clinical response to AJ1-11095 evaluated by spleen volume assessments. | Baseline through Week 24
  Spleen volume reduction (SVR) of ≥35% from Baseline measured by magnetic resonance imaging (MRI) or computed tomography (CT).
To assess clinical response to AJ1-11095 evaluated by spleen length assessments. | Baseline through Week 24
  Proportion of subjects with ≥50% reduction in length of spleen assessed by palpation.
To assess clinical response to AJ1-11095 evaluated through spleen size improvement. | Baseline through Week 24
  Time to spleen size improvement response measured by patient and across all patients.
To evaluate the Area Under the Curve (AUC) of AJ1-11095 | Pre dose and post dose Cycle 1 (Day 1, and Day 2 (24hrs post), Day 8, 15, 22, and Cycle 2 (Day 1 and 24 hrs post).
  AUC time curve from 0 to 24 hrs post dose and percent difference between intervals will be evaluated.
To evaluate the Cmax of AJ1-11095 | Pre dose and post dose Cycle 1 (Day 1, and Day 2 (24hrs post), Day 8, 15, 22, and Cycle 2 (Day 1 and 24 hrs post).
  The maximum observed plasma concentration will be evaluated.
To evaluate the Tmax of AJ1-11095 | Pre dose and post dose Cycle 1 (Day 1, and Day 2 (24hrs post), Day 8, 15, 22, and Cycle 2 (Day 1 and 24 hrs post).
  The duration of time taken to reach Cmax will be evaluated.
To evaluate the half-life of AJ1-11095 | Pre dose and post dose Cycle 1 (Day 1, and Day 2 (24hrs post), Day 8, 15, 22, and Cycle 2 (Day 1 and 24 hrs post).
  The depletion of AJ1-00195 in the body will be observed over time.

CONTACTS AND LOCATIONS:
Overall Officials: John Mascarenhas, M.D., Principal Investigator — Mt. Sinai
Locations (13):
- United States (13):
  - Stanford Cancer Institute, Palo Alto, California
  - Moffitt Cancer Cancer Center, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No